CLINICAL TRIAL: NCT03856762
Title: Dietary Pattern and Metabolic Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAS-HDP-201902
Record Dates: First submitted 2019-02-21; First posted 2019-02-27 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Diet; PreDiabetes; Weight Loss
MeSH Terms: conditions — Prediabetic State; Weight Loss | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional Jiangnan diet (Experimental): Subjects will be supplied with traditional Jiangnan diet and APP-based behavioral modification
  Interventions: Dietary Supplement: traditional Jiangnan diet
- Mediterranean diet (Experimental): Subjects will be supplied with Mediterranean diet and APP-based behavioral modification
  Interventions: Dietary Supplement: Mediterranean diet
- Current Shanghai diet (Experimental): Subjects will be supplied with current Shanghai diet and APP-based behavioral modification
  Interventions: Dietary Supplement: Current Shanghai diet

INTERVENTIONS:
Dietary Supplement: traditional Jiangnan diet — traditional Jiangnan diet supplement from Monday to Friday for six months
  Arms: Traditional Jiangnan diet
Dietary Supplement: Mediterranean diet — Mediterranean diet supplement from Monday to Friday for six months
  Arms: Mediterranean diet
Dietary Supplement: Current Shanghai diet — current Shanghai diet supplement from Monday to Friday for six months
  Arms: Current Shanghai diet

SUMMARY:
This is a single-blind, randomized trial. Based on inclusion and exclusion criteria, 253 eligible volunteers, who were 25-60 years old, with overweight/obese and prediabetes are assigned to one of three dietary patterns: healthy Jiangnan, restricted-calorie; Mediterranean, restricted-calorie; or typical Shanghai, restricted-calorie.

The Shanghai Institutes for Biological Sciences of the Chinese Academy of Sciences(CAS) cooperated with Ruijin Hospital to conduct the study which is funded by the CAS. The study' protocol has been approved by the Ethics Committee of Shanghai Institutes for Biological Sciences. The main purpose of this study is to clarify: the efficacy of traditional Jiangnan dietary pattern, Mediterranean dietary pattern and the current Shanghai dietary pattern in improving overweight/obesity, glucose homeostasis, other cardiovascular metabolic risk factors and their main regulatory factors in Chinese.

DETAILED DESCRIPTION:
Nowadays, the prevalence of type 2 diabetes and its related metabolic diseases is rapidly rising in China. Obesity and early pathoglycemia will increase the risk of diabetes and related cardiovascular diseases severely. Therefore, more effective methods and strategies need to be found to reduce body weight, improve pathoglycemia, and control the development of this high-risk group to type 2 diabetes. As the most popular healthy dietary pattern in the world, the role of Mediterranean diet in the prevention of type 2 diabetes remains unclear. In addition, the protective role of Chinese traditional dietary pattern with lots of plant-based foods in the region of Jiangnan has not been clarified through intervention studies. Therefore, it is urgent to explore the feasibility and effectiveness of traditional Jiangnan diet and Mediterranean diet through dietary intervention studies in Chinese.

The effectiveness of healthy dietary patterns can be further enhanced by limiting dietary intake to achieve weight loss. Recently, the Spainish study found that energy-restricted Mediterranean diet + physical activity + behavioral interventions are more conducive to weight loss in overweight/obesity with prediabetes/type 2 diabetes compared with conventional Mediterranean dietary interventions. The 2019 Diabetes Management Standard of American Diabetes Association re-emphasizes the importance of moderate weight loss for delaying the progression of type 2 diabetes, and recommends that a reduction in dietary intake is 500-750 kcal/day to reach 1-2 pounds per week is suitable. At the same time, the American Clinical Endocrine Society and the American Endocrine Society have also updated the 2019 Comprehensive Management Guide for Type 2 Diabetes. The new guidelines point out that all overweight or obese patients with prediabetes or type 2 diabetes should pay attention to weight loss. And weight loss treatment should include specific lifestyle interventions, including calorie-restricted healthy dietary plan, physical activity and behavioral interventions.

Dietary intervention studies in the past mainly relied on dietary education. However, this study now provides a healthy and reasonable dietary model for the Chinese population through lifestyle intervention to clarify the improvement of cardiovascular metabolic risk such as overweight/obesity, glucose homeostasis, and the scientific basis for establishing a healthy dietary model which is suitable for Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 to 60 years old
* 24.0 ≤ BMI ≤ 40.0 kg/m2
* fasting glucose≥5.6 mmol/L

Exclusion Criteria:

* Diabetes or use of insulin or other hypoglycemic medications
* Pregnancy or lactation
* Trying to change body weight in the way
* Use of antibiotic in the preceding 3 months for 3-serial days
* Obvious changes of medication in the preceding 3 months
* History of drug or alcohol abuse or other substance abuse; (Alcohol abuse is defined as regular alcohol consumption > 40 g/day)
* Any severe liver or renal diseases
* Severe gastrointestinal diseases
* Surgical events preceding 1 year (except appendicitis or hernia surgery)
* Severe cardiovascular or cerebrovascular diseases or phase three hypertension
* Implantation of heart stent
* Cancer or receiving radiotherapy and chemotherapy within 5 years
* Hyperthyroidism or hypothyroidism
* Suffering from hepatitis B, tuberculosis, AIDS and other infectious diseases
* Any mental disorders or current use of antidepressants
* Food contraindications or allergies to foods included in the intervention
* Cognitive disability
* Participated in any other clinical studies within 3 months

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 253 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Body weight | 6 months
  Body weight will be assessed by electronic scale (Seca-882; ScalesGalore) during each visit and Wi-Fi scale at home
Glucose homeostasis | 6 months
  Glucose homeostasis will be assessed by Continuous Glucose Monitoring(FreeStyle Libre)
Glucose | 6 months
  Glucose will be assessed by oral glucose tolerance test

SECONDARY OUTCOMES:
Abdominal fat | 6 months
  Abdominal fat will be assessed using Magnetic Resonance Imaging
Blood pressure | 6 months
  Both systolic pressure and diastolic pressure will be assessed using electronic blood pressure monitor (Omron HEM-7000)
Total cholesterol | 6 months
  Total cholesterol will be assessed using an automatic biochemical analyzer
Triglyceride | 6 months
  Triglyceride will be assessed using an automatic biochemical analyzer
LDL-C | 6 months
  LDL-C will be assessed using an automatic biochemical analyzer
HDL-C | 6 months
  HDL-C will be assessed using an automatic biochemical analyzer
HbA1c | 6 months
  HbA1c will be assessed using liquid Chromatograph Mass Spectrometer

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, PhD, Principal Investigator — Shanghai Institute of Nutrition and Health, Chinese Acadamy of Sciences
Locations (1):
- Ruijin hospital; SAIC FAW-Volkswagen Automobile Co, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ni M, Chen Y, Gu W, Zhang Y, Xu M, Gu Y, Chen Y, Zhu Y, Wang X, Luo Y, Xu Y, Lin X, Zeng YA, Liu R, Wang J. Association Between Circulating Gremlin 2 and beta-Cell Function Among Participants With Prediabetes and Type 2 Diabetes. J Diabetes. 2025 Apr;17(4):e70090. doi: 10.1111/1753-0407.70090. PMID 40270326
- [Derived] Lin H, Wang Q, Gao A, Sun Y, Shen C, Chen Y, Wang Z, Xu X, Ni M, Chen Y, Zhang J, Luo Y, Lin X, Bi Y, Ning G, Wang W, Hong J, Gu W, Wang J, Liu R. Enteropancreatic hormone changes in caloric-restricted diet interventions associate with post-intervention weight maintenance. Clin Nutr. 2024 Dec;43(12):5-14. doi: 10.1016/j.clnu.2024.10.004. Epub 2024 Oct 5. PMID 39418916
- [Derived] Luo Y, Wang J, Sun L, Gu W, Zong G, Song B, Shen C, Zhou P, Chen Y, Wu Y, Lin H, Zheng H, Ni M, Yang X, Chen Y, Xu X, Zhang J, Shi J, Zhang R, Hu J, Hou H, Lu L, Xu X, Liang L, Liu R, Liu X, Li H, Hong J, Wang W, Lin X, Ning G. Isocaloric-restricted Mediterranean Diet and Chinese Diets High or Low in Plants in Adults With Prediabetes. J Clin Endocrinol Metab. 2022 Jul 14;107(8):2216-2227. doi: 10.1210/clinem/dgac303. PMID 35579171